CLINICAL TRIAL: NCT05967455
Title: Phase One, Open Label, Homologous Reinfection With Dengue-1-Virus-Live Virus Human Challenge - (DENV-1-LVHC) or Dengue-3-Virus-Live Virus Human Challenge (DENV-3-LVHC) Virus Strains
Brief Title: Homologous Re-infection With Dengue 1 or Dengue 3
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency); Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2023-01-UMU
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-10

CONDITIONS: Dengue
Keywords: Dengue; Flavivirus Infections; Virus Diseases
MeSH Terms: conditions — Dengue; Flavivirus Infections; Virus Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1 Naive DENV1 (Experimental): Dengue-1-Virus-Live-Virus-Human-Challenge (DENV-1-LVHC), two doses (0.5 mL of 6.5 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously on day 1 and day 181.
  Interventions: Biological: Dengue virus 1 Live Virus Human Challenge (DENV-1-LVHC)
- Cohort 2 Naive DENV3 (Experimental): Dengue-3-Virus-Live-Virus-Human-Challenge (DENV-3-LVHC), two doses (0.5 mL of 1.4 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously on day 1 and day 181.
  Interventions: Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC)
- Cohort 3 Returning DENV1 (Experimental): Dengue-1-Virus-Live-Virus-Human-Challenge (DENV-1-LVHC), single dose (0.5 mL of 6.5 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously on day 1.
  Interventions: Biological: Dengue virus 1 Live Virus Human Challenge (DENV-1-LVHC)
- Cohort 4 Returning DENV3 (Experimental): Dengue-3-Virus-Live-Virus-Human-Challenge (DENV-3-LVHC), single dose (0.5 mL of 1.4 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously on day 1.
  Interventions: Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC)

INTERVENTIONS:
Biological: Dengue virus 1 Live Virus Human Challenge (DENV-1-LVHC) — Dengue subtype 1 Challenge Virus (DENV-1) strain 45AZ5
  Arms: Cohort 1 Naive DENV1; Cohort 3 Returning DENV1
Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC) — Dengue subtype 3 Challenge Virus (DENV-3) strain CH53489
  Arms: Cohort 2 Naive DENV3; Cohort 4 Returning DENV3

SUMMARY:
Previous studies with one dengue infection in a controlled environment at Upstate generated data that has been important in understanding the clinical signs and symptoms and how a person's body reacts to dengue infection over time. This has helped investigators compare what is seen in the clinic to what is seen in areas where dengue is prevalent. The investigators want to collect similar information when a person gets the same dengue twice in a controlled environment with the hope that this will lead them to a better understanding of the disease.

New participants

* will receive one inoculation of dengue and then return to the clinic or be contacted by phone over 6 months;
* will receive a second inoculation after 6 months and return to the clinic or be contacted by phone for three more months;
* will collect saliva at home;
* will allow the study team to collect blood and saliva at the clinic visits.

Participants who have been in previous dengue inoculation studies at SUNY Upstate

* will receive one inoculation of dengue and then return to the clinic or be contacted by phone over 6 months;
* will collect saliva at home;
* will allow the study team to collect blood and saliva at the clinic visits.

All participants will be seen in the clinic every other day for the first three weeks after any inoculation.

DETAILED DESCRIPTION:
The purpose of this study is to explore the clinical, virologic, and immunologic response of subjects following primary controlled dengue infection or following controlled homologous dengue reinfection.

SUNY Upstate Medical University completed three Dengue Human Infection Model studies, two with dengue 1 (DENV-1-LVHC), NCT 02372175 and NCT 03869060, and one with dengue 3 (DENV-3-LVHC), NCT 04298138 and investigators gained incredible knowledge about primary dengue infection. The investigators are moving to the next step in acquiring knowledge about the kinetics of homologous secondary infection in a controlled setting in this study. People who acquire natural dengue infection and who are subsequently infected by the same serotype are thought to have lifelong protection to that serotype.

Investigators will recruit up to 10 naive participants and infect them with either DENV-1-LVHC or DENV-3-LVHC with the same dose of virus as in previous studies. These participants will be followed over 6 months and reinfected with the same serotype originally received, i.e. homologous reinfection, and followed for another three months. Investigators will also recruit up to 10 participants who received either DENV-1-LVHC or DENV-3-LVHC in previous studies. These participants will be reinfected with the same serotype that was previously received and followed for 6 months. Investigators intend to collect similar information about the kinetics of homologous secondary infection as was collected in the studies following primary infection.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-55 at the time of consent
2. Ability and willingness to sign informed consent
3. Passing score on comprehension test of at least 75%, with up to 3 attempts
4. Available for the study period
5. Willing to use contraception for the duration of the study (birth control pills or patches, intrauterine device (IUD), Depo-Provera, implantable birth control (implants of levonorgestrel), estrogenic vaginal ring, tubal ligation, vasectomy of the sole male partner, male condom combined with a vaginal spermicide (foam, gel, film, cream, or suppository), male condom combined with a female diaphragm, either with or without vaginal spermicide, partner in a homosexual relationship, abstinence)
6. Provide consent for release of medical history records from primary care physician, college or university, urgent care or emergency room visit

Exclusion Criteria:

1. Female: pregnant or lactating
2. Heavy menstrual bleeding within the last 6 months- menstrual periods lasting longer than 6 days or requiring 5 or more pads or tampons per day, endometriosis or uterine scarring
3. Women who intend to become pregnant or men who intend to father a child during the study period (approximately 209 days for Cohorts 1 and 2 and approximately 91 days for Cohorts 3 and 4)
4. Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B (assessed by HbsAg) virus
5. Positive antibodies to dengue (cohorts 1 and 2). If the subject has previously screened negative for dengue in the last 12 months and has not traveled to an endemic area. The results of the previous screening will be used.
6. Any history of dengue infection or dengue vaccination (licensed or experimental) (cohorts 1 and 2); or planned dengue vaccination during the study period (all cohorts)
7. Recent (in the past 4 weeks) travel to any dengue endemic area or travel to a country with risk of yellow fever or Japanese encephalitis transmission
8. Positive urine screen for cocaine, amphetamines, opiates or methadone
9. Currently taking anti-coagulant medication, aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
10. Active diabetes, active peptic ulcer disease (PUD), chronic obstructive pulmonary disease (COPD), coronary artery disease (CAD)
11. Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
12. Current, or a history of, auto-immune disease other than well controlled Hashimoto's thyroiditis
13. History of Guillain-Barré syndrome (GBS)
14. Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the subject from participating in the study.
15. Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous vaccination or an allergy to specific medications/animals for which antigens may be in the virus preparations to include: shellfish allergy, fetal bovine serum, L-glutamine, neomycin and streptomycin
16. Chronic migraine headaches, defined as more than 15 headache days per month over a 3 month period of which more than 8 are migraines, in the absence of medication over use
17. Planning to donate blood in the 1 year following inoculation with dengue
18. Recent blood donation within prior 14 days of inoculation
19. Receipt of blood products or antibodies within 56 days of inoculation or during the study period
20. Planned travel during the study period (approximately 210 days for Cohorts 1 and 2 and approximately 91 days for Cohorts 3 and 4) which would interfere with the ability to complete all study visits
21. Subjects with the following grade 2 or greater lab abnormalities: Creatinine; ALT, AST; Hemoglobin (females and males); WBC; Platelets; PT; PTT; Fibrinogen
22. Any laboratory abnormalities prior to inoculation that are considered by the investigator to be clinically significant in addition those listed above
23. Significant screening physical examination abnormalities or chronic medical condition that in the opinion of the investigator may impact subject safety
24. Participation (active or follow-up phase) or planned participation in another vaccine, drug, or medical device in the 4 weeks prior to this trial or during the trial
25. Recent or scheduled receipt of any vaccine 4 weeks prior to or after virus inoculation
26. Beliefs that bar the administration of blood products or transfusions
27. Clinician discretion

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-08-26 (Actual); Study Completion 2024-08-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of Solicited Injection Site Symptoms | 6 days post virus inoculation
  Number of solicited symptoms
Intensity of Solicited Injection Site Symptoms | 6 days post virus inoculation
  Graded according to FDA Tables for Clinical Abnormalities: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe), Grade 4 (Potentially life threatening)
Duration of Solicited Injection Site Symptoms | 6 days post virus inoculation
  Number of days per symptom
Occurrence of Solicited Systemic Symptoms | 20 day post primary infection for cohorts 1 and 2 and 20 days post reinfection, all cohorts
  Number of solicited symptoms
Intensity of Solicited Systemic Symptoms | 20 day post primary infection, cohorts 1 and 2 and 20 days post reinfection, all cohorts
  Graded according to FDA Tables for Clinical Abnormalities: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe), Grade 4 (Potentially life threatening)
Duration of Solicited Systemic Symptoms | 20 day post primary infection, cohorts 1 and 2 and 20 days post reinfection, all cohorts
  Number of days per symptom
Occurrence of Unsolicited Systemic Symptoms | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Number of unsolicited symptom
Intensity of Unsolicited Systemic Symptoms | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Graded according to FDA Tables for Clinical Abnormalities: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe), Grade 4 (Potentially life threatening)
Duration of Unsolicited Systemic Symptoms | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Number of days per symptom
Number of Abnormal Laboratory Measurements | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Total number of all abnormal labs
Intensity of Abnormal Laboratory Measurements | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Graded according to SUNY Upstate clinical laboratory normals and FDA Tables for Laboratory Abnormalities: Grade 1 (Mild), Grade 2 (Moderate), Grade 3 (severe), Grade 4 (Potentially life threatening)
Duration of Abnormal Laboratory Measurements | 28 day post primary infection, cohorts 1 and 2 and 28 days post reinfection, all cohorts
  Number of days of abnormal labs
Number of Serious Adverse Events | 6 months post primary infection, cohorts 1 and 2
  Total number
Number of Serious Adverse Events | 3 months post reinfection, cohorts 1 and 2
  Total number
Number of Serious Adverse Events | 6 months post reinfection, cohorts 3 and 4
  Total number

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Thomas, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- State University of New York, Upstate Medical University (SUNY-UMU), Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Endy TP, Wang D, Polhemus ME, Jarman RG, Jasper LE, Gromowski G, Lin L, De La Barra RA, Friberg H, Currier JR, Abbott M, Ware L, Klick M, Paolino KM, Blair DC, Eckels K, Rutvisuttinunt W, Thomas SJ. A Phase 1, Open-Label Assessment of a Dengue Virus-1 Live Virus Human Challenge Strain. J Infect Dis. 2021 Feb 3;223(2):258-267. doi: 10.1093/infdis/jiaa351. PMID 32572470
- [Result] Waickman AT, Lu JQ, Fang H, Waldran MJ, Gebo C, Currier JR, Ware L, Van Wesenbeeck L, Verpoorten N, Lenz O, Tambuyzer L, Herrera-Taracena G, Van Loock M, Endy TP, Thomas SJ. Evolution of inflammation and immunity in a dengue virus 1 human infection model. Sci Transl Med. 2022 Oct 26;14(668):eabo5019. doi: 10.1126/scitranslmed.abo5019. Epub 2022 Oct 26. PMID 36288280